CLINICAL TRIAL: NCT02070055
Title: Dietary Correlates of the Maximal Capacity for Fat Oxidation During Exercise in Males and Females.
Brief Title: Dietary Correlates of the Maximal Capacity for Fat Oxidation
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Gareth Fletcher, Doctoral Researcher, University of Birmingham
Other Study IDs: RG_12-251
Record Dates: First submitted 2012-12-06; First posted 2014-02-24 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Maximal Rate of Fat Oxidation
Keywords: Maximal Rate of Fat Oxidation; Substrate Oxidation; Fat oxidation; Respiratory Exchange Ratio (RER); Exercise; indirect calorimetry; substrate crossover
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment: No treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
There is a large variability in people's ability to burn fat during exercise. It is thought that differences in dietary intake can partly explain this variation, however this has not been comprehensively studied. This will be investigated by measuring participant's habitual diet and rates of fat oxidation during exercise, and look for associations between the two.

DETAILED DESCRIPTION:
The capacity to oxidize (burn) fat as fuel for exercise may have important implications for health and performance. For example, increased fat oxidation could help to induce a negative fat balance and over time improve body composition. Furthermore, increasing the oxidation of fat could spare carbohydrate utilization during exercise which should improve endurance performance by preserving the bodies limited carbohydrate reserves for the latter stages of competition. Interestingly, there is substantial individual variation in the balance of fuels used for energy during exercise and in particular the maximal capacity to oxidize fat (MFO). Whilst habitual diet is known to affect the metabolic response to exercise, the influence of nutrition on the individual variability observed in maximal fat oxidation has not been comprehensively studied.

Therefore, the proposed investigation aims to build on current understanding of how various nutritional factors influence MFO during exercise. Based on previous small intervention studies, it is suspected that energy balance and macronutrient content or distribution may exert the strongest influence on MFO during exercise. Specifically, the main hypothesis would be that negative energy balance; higher fat intake and/or low carbohydrate intake would be the strongest positive influencer's of MFO. Nonetheless, the determination of an array of habitual and acute nutrient intake data in a relatively large cohort of healthy individuals will enable an insight into the influence of a comprehensive array of nutrients on MFO during exercise. With a greater understanding of the nutritional factors that influence MFO during exercise, new nutritional interventions can be designed to promote the oxidation of fat for improved health and performance.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 45 years of age
2. Sex: Men and women*

   * Women must be eumenorrheic and regularly menstruating or using hormonal contraception
3. BMI: 18.8-29.9 kg/m2
4. Diagnosis / General Health: Good general health and accustomed to normal levels of activity as assessed by the School of Sport and Exercise Sciences General Health Questionnaire
5. Compliance: understands and is willing, able and likely to comply with all study procedures and restrictions.
6. Consent: demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.

Exclusion Criteria:

1. Women who are known to be pregnant
2. Women who are breast feeding
3. Current or recent (last 3 months) participation in another clinical or intervention trial.
4. Concomitant Medication. Prescription or non-prescription medication that may interfere with metabolism or substrate utilisation (including beta-blockers, insulin, bronchodilators, anti-inflammatory agents, thyroxine and medications/supplements that in the opinion of the investigator may affect metabolism).
5. Substance abuse (within the last 1 years)
6. Completely sedentary individuals as assessed by the School of Sport and Exercise Sciences General Health Questionnaire
7. Consumption of alcohol 24 hours prior to Visit 2
8. Current or recent (within the last 30 days) smoker
9. Engaged in prolonged periods of food abstinence (e.g., for health or religious reasons) that may influence the normal metabolic response to exercise

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Local healthy population
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Rate of Maximal Fat Oxidation in grams per minute | From any 10 second interval from a 30 minute exercise test
  To determine the extent to which the habitual diet influences the maximal rate of fat oxidation during exercise in healthy men and women

CONTACTS AND LOCATIONS:
Overall Officials: Gareth A Wallis, Dr, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Fletcher G, Eves FF, Glover EI, Robinson SL, Vernooij CA, Thompson JL, Wallis GA. Dietary intake is independently associated with the maximal capacity for fat oxidation during exercise. Am J Clin Nutr. 2017 Apr;105(4):864-872. doi: 10.3945/ajcn.116.133520. Epub 2017 Mar 1. PMID 28251936